CLINICAL TRIAL: NCT07305480
Title: Longitudinal Observational Study for Developing and Validating a Digital Twin Model of Human Blastocyst Development, Implantation Potential, and Pregnancy Outcomes Using Fully De-Identified, Multimodal IVF Clinical and Molecular Data
Brief Title: Longitudinal Clinical Observation of a Digital Twin Model for Blastocyst Evaluation in IVF Clinics
Acronym: IVFDT
Status: Active, not recruiting | Type: Observational
Sponsor: Ukraine Association of Biobank (Other)
Responsible Party: Sponsor
Other Study IDs: IVFDT-LONGOBS-001; UABA-IVF-DT-001 (Registry Identifier: Ukrainian Association of Biobanks Austria (UABA) - Digital Twin IVF Registry)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Implantation, Embryo
Keywords: IVF; Digital Twin; Embryo selection; Multi-omics; Pregnancy outcomes; AI modeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: IVF Patients Monitored With Digital Twin Embryo Evaluation: This cohort includes patients undergoing in-vitro fertilization (IVF) whose embryos are evaluated using the Digital Twin model for blastocyst quality and implantation prediction. No clinical intervention is performed. The study collects multi-omics, morphological, and clinical data to monitor implantation success, pregnancy progression, and neonatal outcomes up to 3 years after birth.
  Interventions: Other: Digital Twin Computational Modeling

INTERVENTIONS:
Other: Digital Twin Computational Modeling — Computational digital twin model that analyzes fully de-identified, non-image clinical, molecular, biochemical, and laboratory data from routine IVF care to evaluate embryo implantation potential. The model does not influence clinical decision-making and is used only for retrospective and prospective observational analysis.

SUMMARY:
This study aims to develop and validate a non-image, multimodal digital twin model of the human blastocyst using fully de-identified clinical, laboratory, molecular, biochemical, and long-term follow-up data obtained during routine IVF treatment. The dataset includes parental clinical background, IVF cycle parameters, embryo morphology in text format, PGT-A results, secretome and exosomal biomarkers, endometrial receptivity profiles, pregnancy course, delivery outcomes, and child development data up to 3 years of age.

The purpose of this observational study is to create a longitudinal reference dataset linking embryo-level molecular and biochemical characteristics with clinical outcomes from implantation to early childhood. The digital twin model is intended to investigate predictors of implantation success, embryo viability, and early developmental trajectories without the use of images or videos. No investigational drugs or devices are used, and no procedures beyond standard clinical practice are added.

DETAILED DESCRIPTION:
This observational study collects and integrates multimodal, non-image data from routine IVF cycles to construct digital twin models of human blastocysts. The dataset includes synchronized molecular, cellular, biochemical, and clinical parameters describing both the embryo and the maternal environment during implantation and early pregnancy. All information is fully de-identified and obtained as part of standard clinical care.

Parental and Clinical Background

The dataset incorporates:

demographic factors, reproductive history, and relevant risk factors;

karyotype results, thrombophilia and autoimmune screening;

sperm DNA fragmentation indices;

ovarian stimulation parameters and hormonal dynamics throughout the IVF cycle.

IVF Laboratory Data

Non-image embryologic information includes:

oocyte maturity and fertilization method (e.g., ICSI);

early cleavage development documented in descriptive text format (no images or videos);

blastocyst grading;

preimplantation genetic testing for aneuploidy (PGT-A), including ploidy status and mosaicism.

Molecular and Secretome Data

Embryo- and culture-media-associated biomarkers include:

cytokines, growth factors, LIF, and metabolic indicators in spent media;

exosomal microRNA signatures linked to implantation potential;

transcriptomic and methylation profiles of trophectoderm samples when available.

Endometrial and Immune Environment

Maternal environment assessment includes:

transcriptomic profiling of the endometrial receptivity window (ERA-like signatures);

uterine immune parameters such as uNK cell activity and T-regulatory balance.

Pregnancy, Delivery, and Child Follow-Up

Collected follow-up information includes:

β-hCG kinetics, early ultrasound development, and pregnancy complications;

delivery outcomes and newborn characteristics;

longitudinal developmental assessments of the child up to 3 years of age.

Study Objectives

To construct digital twin representations of individual blastocysts by integrating multi-omics and clinical parameters obtained during IVF.

To identify non-invasive biomarkers of implantation success and embryo viability.

To analyze associations between early embryo molecular profiles and neonatal or early childhood developmental outcomes.

Study Design

This is a non-interventional, observational study. All data are obtained retrospectively and/or prospectively from routine clinical practice in IVF clinics. No experimental procedures, investigational drugs, or investigational devices are introduced. Participation involves only the use of fully de-identified clinical, laboratory, and follow-up data for research purposes. Parents provide informed consent for use of de-identified information.

The study is not conducted under an IND or IDE, and it does not involve FDA-regulated products.

Significance

The resulting longitudinal dataset will support the development of AI-based digital twin models, facilitate biomarker discovery, and advance precision reproductive medicine. These models aim to predict blastocyst competence, implantation potential, and early developmental trajectories using non-image, multimodal clinical and molecular data.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing in vitro fertilization (IVF) treatment at participating fertility clinics.
* Availability of non-image embryo development data.
* Availability of text-based morphological embryo descriptions.
* Availability of PGT-A results.
* Availability of secretome and exosomal biomarker data.
* Availability of molecular and biochemical data collected during routine clinical care.
* Availability of IVF cycle parameters collected during routine clinical workflow.
* Embryos evaluated according to standard clinic protocols with documented implantation outcomes.
* Age of the oocyte provider between 20 and 42 years.
* Signed informed consent allowing use of fully de-identified clinical, laboratory, molecular, and follow-up data.

Exclusion Criteria:

* Embryos lacking sufficient non-image developmental data required for digital twin generation or implantation outcome assessment.
* Use of donor oocytes or donor embryos when linkage with required clinical or laboratory metadata is not possible.
* Cases in which implantation outcome cannot be confirmed.
* Presence of severe uterine abnormalities prior to embryo transfer that may affect implantation reliability.
* Withdrawal of consent for use of anonymized clinical, laboratory, or follow-up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes women undergoing in vitro fertilization (IVF) treatment whose embryo-related clinical, laboratory, molecular, and biochemical data are collected as part of routine clinical care. The dataset consists of fully de-identified non-image embryo development information, including text-based morphological descriptions, PGT-A results, secretome and exosomal biomarkers, endometrial receptivity profiles, and IVF cycle parameters required to construct and validate a multimodal digital twin model of blastocyst implantation potential.
  Participants represent typical reproductive-age IVF patients receiving standard ovarian stimulation, oocyte retrieval, embryo culture, assessment, and embryo transfer procedures. No experimental interventions, investigational drugs, or investigational devices are used. Only retrospective and/or prospectively collected routine clinical data are analyzed for computational model development.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Digital Twin Model in Predicting Embryo Implantation | From embryo transfer (Day 0) to confirmation of clinical pregnancy (up to 12 weeks of gestation).
  Evaluation of the predictive performance of the digital twin model for embryo implantation outcomes based on integrated multi-omics, morphokinetic, and clinical data. The accuracy will be measured by AUC, sensitivity, specificity, and calibration metrics against real clinical implantation outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ukrainian Association of Biobanks Austria - Digital Twin Lab, Graz, Austria

IPD SHARING:
Plan to Share IPD: No